CLINICAL TRIAL: NCT03052036
Title: The British Heart Foundation Older Patients With Non-ST SEgmeNt elevatIOn myocaRdial Infarction Randomized Interventional TreAtment Trial
Brief Title: The British Heart Foundation SENIOR-RITA Trial
Acronym: SENIOR-RITA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: British Heart Foundation (Other); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7910
Record Dates: First submitted 2017-01-11; First posted 2017-02-14 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI
Keywords: Acute Coronary Syndrome
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Invasive Treatment (Other): Coronary angiography with a view to coronary revascularisation
  Interventions: Procedure: Coronary Angiography; Procedure: Coronary revascularisation; Other: Optimal Medical Therapy
- Optimal Medical Therapy (Other): Patients to be treated with guideline recommended secondary prevention therapy including antiplatelet therapy, statins, ACE inhibitors, betabloackers
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Procedure: Coronary Angiography — Coronary angiography to determine location of blocked or narrowed arteries.
  Arms: Invasive Treatment
Procedure: Coronary revascularisation — PCI or CABG will be performed following coronary angiography at the discretion of the treating cardiologist.
  Arms: Invasive Treatment
Other: Optimal Medical Therapy — Patients to receive conservative treatment in the form of guideline recommended secondary prevention therapy including antiplatelet therapy, statins, ACE Inhibitors and beta blockers.

SUMMARY:
SENIOR-RITA is a multicentre prospective open-label trial randomizing patients presenting with type 1 NSTEMI aged ≥75 years between invasive and conservative treatment strategies, to compare time from randomisation to cardiovascular death or non-fatal MI

DETAILED DESCRIPTION:
The population is getting older and heart artery disease is the biggest killer in the UK. Over recent years, there have been improvements in medications and technologies to treat it, but these have been primarily tested in younger patients. Previous research studies suggest that older patients (75 years and over) are not well represented in clinical research and these patients in particular those that are frail and those with co-morbidities are less likely to receive advanced medications and medical procedures. The current study will enrol patients 75 years and over, presenting with a heart attack. If patients agree to participate, they will be randomly allocated to one of two treatment groups. In the first group, patients will receive the latest medications recommended in heart attack. In the second group, in addition to these medications, patients will have coronary angiography. This will show whether they have any blockages in heart arteries. If appropriate, coronary revascularisation by percutaneous coronary intervention (PCI) commonly known as coronary angioplasty or coronary artery bypass grafting, sometimes called CABG (a surgical procedure in which a blood vessel from the leg, arm or chest is used to bypass a narrowed section of a coronary artery) will be carried out. During the trial, frailty scores, cognition measures, co-morbidity indices, questionnaires on quality of life, NHS and personal social services utilization will be collected from the participant and in addition proxy quality of life information will be collected from the participant's carers. Investigators will evaluate which one of the two treatment groups will do better and live longer. Investigators will also collect information on their quality of life and frailty measures for a 5 year period. The trial hopes to recruit 2300 patients from approximately 30 centres across the UK.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 75 years
* Type 1 NSTEMI during index hospitalisation

Exclusion Criteria:

* Patients presenting with STEMI or unstable angina
* Patients with cardiogenic shock
* Patients with known life expectancy <1 year
* Patients in whom neither the patient nor the consultee are able and willing to provide written informed consent
* Previous inclusion in the BHF SENIOR-RITA trial
* Inability to undergo invasive coronary angiography, such as no vascular access site, or absolute contraindication to coronary revascularisation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1518 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Time to cardiovascular death or non-fatal MI (defined by the fourth universal definition) from randomization | Up to 5 years
  To determine the impact of a routine invasive strategy on cardiovascular death and non-fatal myocardial infarction (MI) compared with a conservative treatment strategy in older patients (≥75 years) with NSTEMI.

SECONDARY OUTCOMES:
All cause, cardiovascular and non-cardiovascular death rates | Up to 5 years
Recurrent myocardial infarction | Up to 5 years
Hospitalisation for heart failure | Up to 5 years
Urgent coronary revascularisation | Up to 5 years
Recurrent hospitalisation for myocardial infarction | Up to 5 years
Stroke | Up to 5 years
Length of time spent at home | Up to 5 years
Fried and Rockwood frailty scores | Up to 5 years
Quality of Life using EQ-5D-5L and quality adjusted life years (QALY) | Up to 5 years
  Quality of life will be measured using the EQ-5D-5L instrument[REF: The EuroQol Group (1990). EuroQol-a new facility for the measurement of health-related quality of life. Health Policy 16(3):199-208html ] (paper and telephone versions), with the results for each participant converted into quality-adjusted life-years (QALYs) using the area under the curve approach, a standard methodology for this process,[REF: Drummond MOB, B; Stoddart, G; Torrance, G. . Methods for the economic evaluation of Health Care Programmes: Oxford University Press 2005.] with the responses to the EQ-5D-5L scored using the appropriate value set for the United Kingdom, which is expected to be available by the time of the analysis. REF: Office for Health Economics. New OHE Publications: An EQ-5D-5L Value Set for England. Available at: https://www.ohe.org/news/new-ohe-publications-eq-5d-5l-value-set-england. Accessed February 03 2017]
Costs to the NHS and personal social services | Up to 5 years
Incremental cost per QALY gained at 1 year | Up to 5 years
Procedural complications | Within 7 days of invasive care
  Perforation, myocardial infarction (Type 4a), coronary dissection, TIA, Death in Cath Lab, Aortic dissection
Bleeding | Up to 1 year
  Bleeding according to BARC Criteria
Renal replacement therapy | Within 7 days of invasive care
  Need for renal replacement therapy
25% increase in serum creatinine concentration | Within 7 days of invasive care
  25% increase in serum creatinine concentration from baseline (hospitalisation)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Vijay Kunadian, MBBS MD FRCP, Principal Investigator — Newcastle University
Locations (40):
- United Kingdom (40):
  - Pinderfields General Hospital, Wakefield, West Yorkshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Basildon & Thurrock University Hospitals NHS Foundation Trust, Basildon
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Broomfield Hospital, Mid Essex Hospitals NHS Trust, Broomfield
  - Cumberland Infirmary, North Cumbria University Hospitals NHS Trust, Carlisle
  - St Helier Hospital, Epsom & St Helier University Hospitals NHS Trust, Carshalton
  - Chesterfield Royal Hospital NHS Foundation Trust, Chesterfield
  - County Durham & Darlington NHS Foundation Trust, Darlington
  - Royal Derby Hospital, Derby Teaching Hospitals NHS Foundation Trust, Derby
  - Ninewells Hospital, NHS Tayside, Dundee
  - Lanarkshire East Kilbride NHS Foundation Trust, East Kilbride
  - East Sussex NHS Healthcare Trust, Eastbourne
  - Royal Infirmary of Edinburgh, Edinburgh
  - Gateshead Hospitals NHS Foundation Trust, Gateshead
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Alexandra Hospital, Glasgow
  - North Tees and Hartlepool Foundation Trust, Hartlepool
  - NHS Ayrshire & Arran, Kilmarnock
  - Leeds General Infirmary, Leeds
  - United Lincolnshire Healthcare Trust, Lincoln
  - London Royal Free, Royal Free London NHS Foundation Trust, London
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Chelsea and Westminster, London
  - Wythenshawe Hospital, University Hospital of South Manchester NHS Foundation Trust, Manchester
  - Borders General Hospital, Melrose
  - South Tees NHS Foundation Trust, Middlesbrough
  - The Newcastle Upon Tyne Hospital NHS Foundation Trust, Newcastle upon Tyne
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Pennine Acute Hospitals NHS Trust, Oldham
  - Plymouth Hospital, Plymouth Hospitals NHS Trust, Plymouth
  - Royal Berkshire Hospital, Royal Berkshire Foundation NHS Trust, Reading
  - East Surrey Hospital, Surrey & Sussex NHS Trust, Redhill
  - Salford Royal NHS Foundation Trust, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - South Tyneside NHS Foundation Trust, South Shields
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Torbay Hospital, Torbay & South Devon NHS Foundation Trust, Torquay
  - The York Hospital, York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Orimo H, Ito H, Suzuki T, Araki A, Hosoi T, Sawabe M. Reviewing the definition of "elderly". Geriatrics & Gerontology International. 2006;6:149-158
- [Background] Townsend N, Wickramasinghe K, Bhatnagar P, Smolina K, Nichols M, Leal J, Luengo-Fernandez R, Rayner M. Coronary heart disease statistics 2012 edition. 2012
- [Background] Machin D, Campbell MJ, Tan SB, Tan SH. Comparing survival curves. Sample size tables for clinical studies. Wiley-Blackwell; 2009:84-101.
- [Background] Zaman MJ, Stirling S, Shepstone L, Ryding A, Flather M, Bachmann M, Myint PK. The association between older age and receipt of care and outcomes in patients with acute coronary syndromes: a cohort study of the Myocardial Ischaemia National Audit Project (MINAP). Eur Heart J. 2014 Jun 14;35(23):1551-8. doi: 10.1093/eurheartj/ehu039. Epub 2014 Mar 18. PMID 24644310
- [Background] Beecham J KM. Costing psychiatric interventions. In: Thornicroft, graham, ed. Measuring mental health needs (second edition). Royal college of psychiatrists, london, 2001, 200-224. Measuring Mental Health Needs 2001;Second Edition 24
- [Result] Fox KA, Clayton TC, Damman P, Pocock SJ, de Winter RJ, Tijssen JG, Lagerqvist B, Wallentin L; FIR Collaboration. Long-term outcome of a routine versus selective invasive strategy in patients with non-ST-segment elevation acute coronary syndrome a meta-analysis of individual patient data. J Am Coll Cardiol. 2010 Jun 1;55(22):2435-45. doi: 10.1016/j.jacc.2010.03.007. Epub 2010 Mar 30. PMID 20359842
- [Result] Fox KA, Poole-Wilson PA, Henderson RA, Clayton TC, Chamberlain DA, Shaw TR, Wheatley DJ, Pocock SJ; Randomized Intervention Trial of unstable Angina Investigators. Interventional versus conservative treatment for patients with unstable angina or non-ST-elevation myocardial infarction: the British Heart Foundation RITA 3 randomised trial. Randomized Intervention Trial of unstable Angina. Lancet. 2002 Sep 7;360(9335):743-51. doi: 10.1016/s0140-6736(02)09894-x. PMID 12241831
- [Result] Goodman SG, Huang W, Yan AT, Budaj A, Kennelly BM, Gore JM, Fox KA, Goldberg RJ, Anderson FA Jr; Expanded Global Registry of Acute Coronary Events (GRACE2) Investigators. The expanded Global Registry of Acute Coronary Events: baseline characteristics, management practices, and hospital outcomes of patients with acute coronary syndromes. Am Heart J. 2009 Aug;158(2):193-201.e1-5. doi: 10.1016/j.ahj.2009.06.003. PMID 19619694
- [Result] Devlin G, Gore JM, Elliott J, Wijesinghe N, Eagle KA, Avezum A, Huang W, Brieger D; GRACE Investigators. Management and 6-month outcomes in elderly and very elderly patients with high-risk non-ST-elevation acute coronary syndromes: The Global Registry of Acute Coronary Events. Eur Heart J. 2008 May;29(10):1275-82. doi: 10.1093/eurheartj/ehn124. Epub 2008 Apr 2. PMID 18387940
- [Result] Nguyen HL, Goldberg RJ, Gore JM, Fox KA, Eagle KA, Gurfinkel EP, Spencer FA, Reed G, Quill A, Anderson FA Jr. Age and sex differences, and changing trends, in the use of evidence-based therapies in acute coronary syndromes: perspectives from a multinational registry. Coron Artery Dis. 2010 Sep;21(6):336-44. doi: 10.1097/MCA.0b013e32833ce07c. PMID 20661139
- [Result] Avezum A, Makdisse M, Spencer F, Gore JM, Fox KA, Montalescot G, Eagle KA, White K, Mehta RH, Knobel E, Collet JP; GRACE Investigators. Impact of age on management and outcome of acute coronary syndrome: observations from the Global Registry of Acute Coronary Events (GRACE). Am Heart J. 2005 Jan;149(1):67-73. doi: 10.1016/j.ahj.2004.06.003. PMID 15660036
- [Result] Alexander KP, Newby LK, Cannon CP, Armstrong PW, Gibler WB, Rich MW, Van de Werf F, White HD, Weaver WD, Naylor MD, Gore JM, Krumholz HM, Ohman EM; American Heart Association Council on Clinical Cardiology; Society of Geriatric Cardiology. Acute coronary care in the elderly, part I: Non-ST-segment-elevation acute coronary syndromes: a scientific statement for healthcare professionals from the American Heart Association Council on Clinical Cardiology: in collaboration with the Society of Geriatric Cardiology. Circulation. 2007 May 15;115(19):2549-69. doi: 10.1161/CIRCULATIONAHA.107.182615. PMID 17502590
- [Result] Hordijk-Trion M, Lenzen M, Wijns W, de Jaegere P, Simoons ML, Scholte op Reimer WJ, Bertrand ME, Mercado N, Boersma E; EHS-CR Investigators. Patients enrolled in coronary intervention trials are not representative of patients in clinical practice: results from the Euro Heart Survey on Coronary Revascularization. Eur Heart J. 2006 Mar;27(6):671-8. doi: 10.1093/eurheartj/ehi731. Epub 2006 Jan 19. PMID 16423872
- [Result] Granger CB, Goldberg RJ, Dabbous O, Pieper KS, Eagle KA, Cannon CP, Van De Werf F, Avezum A, Goodman SG, Flather MD, Fox KA; Global Registry of Acute Coronary Events Investigators. Predictors of hospital mortality in the global registry of acute coronary events. Arch Intern Med. 2003 Oct 27;163(19):2345-53. doi: 10.1001/archinte.163.19.2345. PMID 14581255
- [Result] Bagnall AJ, Goodman SG, Fox KA, Yan RT, Gore JM, Cheema AN, Huynh T, Chauret D, Fitchett DH, Langer A, Yan AT; Canadian Acute Coronary Syndrome Registry I and II Investigators; Canadian Global Registry of Acute Coronary Events (GRACE/GRACE2) Investigators. Influence of age on use of cardiac catheterization and associated outcomes in patients with non-ST-elevation acute coronary syndromes. Am J Cardiol. 2009 Jun 1;103(11):1530-6. doi: 10.1016/j.amjcard.2009.01.369. Epub 2009 Apr 8. PMID 19463511
- [Result] Fox KA, Anderson FA Jr, Dabbous OH, Steg PG, Lopez-Sendon J, Van de Werf F, Budaj A, Gurfinkel EP, Goodman SG, Brieger D; GRACE investigators. Intervention in acute coronary syndromes: do patients undergo intervention on the basis of their risk characteristics? The Global Registry of Acute Coronary Events (GRACE). Heart. 2007 Feb;93(2):177-82. doi: 10.1136/hrt.2005.084830. Epub 2006 Jun 6. PMID 16757543
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Result] Ekerstad N, Swahn E, Janzon M, Alfredsson J, Lofmark R, Lindenberger M, Andersson D, Carlsson P. Frailty is independently associated with 1-year mortality for elderly patients with non-ST-segment elevation myocardial infarction. Eur J Prev Cardiol. 2014 Oct;21(10):1216-24. doi: 10.1177/2047487313490257. Epub 2013 May 3. PMID 23644488
- [Result] Ekerstad N, Swahn E, Janzon M, Alfredsson J, Lofmark R, Lindenberger M, Carlsson P. Frailty is independently associated with short-term outcomes for elderly patients with non-ST-segment elevation myocardial infarction. Circulation. 2011 Nov 29;124(22):2397-404. doi: 10.1161/CIRCULATIONAHA.111.025452. Epub 2011 Nov 7. PMID 22064593
- [Result] Veerasamy M, Edwards R, Ford G, Kirkwood T, Newton J, Jones D, Kunadian V. Acute coronary syndrome among older patients: a review. Cardiol Rev. 2015 Jan-Feb;23(1):26-32. doi: 10.1097/CRD.0000000000000016. PMID 24407049
- [Result] Pfisterer M, Buser P, Osswald S, Allemann U, Amann W, Angehrn W, Eeckhout E, Erne P, Estlinbaum W, Kuster G, Moccetti T, Naegeli B, Rickenbacher P; Trial of Invasive versus Medical therapy in Elderly patients (TIME) Investigators. Outcome of elderly patients with chronic symptomatic coronary artery disease with an invasive vs optimized medical treatment strategy: one-year results of the randomized TIME trial. JAMA. 2003 Mar 5;289(9):1117-23. doi: 10.1001/jama.289.9.1117. PMID 12622581
- [Result] Bauer T, Koeth O, Junger C, Heer T, Wienbergen H, Gitt A, Zahn R, Senges J, Zeymer U; Acute Coronary Syndromes Registry (ACOS) Investigators. Effect of an invasive strategy on in-hospital outcome in elderly patients with non-ST-elevation myocardial infarction. Eur Heart J. 2007 Dec;28(23):2873-8. doi: 10.1093/eurheartj/ehm464. Epub 2007 Nov 2. PMID 17982163
- [Result] Savonitto S, Cavallini C, Petronio AS, Murena E, Antonicelli R, Sacco A, Steffenino G, Bonechi F, Mossuti E, Manari A, Tolaro S, Toso A, Daniotti A, Piscione F, Morici N, Cesana BM, Jori MC, De Servi S; Italian Elderly ACS Trial Investigators. Early aggressive versus initially conservative treatment in elderly patients with non-ST-segment elevation acute coronary syndrome: a randomized controlled trial. JACC Cardiovasc Interv. 2012 Sep;5(9):906-16. doi: 10.1016/j.jcin.2012.06.008. PMID 22995877
- [Result] Sinclair H, Kunadian V. Coronary revascularisation in older patients with non-ST elevation acute coronary syndromes. Heart. 2016 Mar;102(6):416-24. doi: 10.1136/heartjnl-2015-307859. Epub 2016 Jan 6. PMID 26740483
- [Result] Lee PY, Alexander KP, Hammill BG, Pasquali SK, Peterson ED. Representation of elderly persons and women in published randomized trials of acute coronary syndromes. JAMA. 2001 Aug 8;286(6):708-13. doi: 10.1001/jama.286.6.708. PMID 11495621
- [Result] Kandzari DE, Roe MT, Chen AY, Lytle BL, Pollack CV Jr, Harrington RA, Ohman EM, Gibler WB, Peterson ED. Influence of clinical trial enrollment on the quality of care and outcomes for patients with non-ST-segment elevation acute coronary syndromes. Am Heart J. 2005 Mar;149(3):474-81. doi: 10.1016/j.ahj.2004.11.014. PMID 15864236
- [Result] Alter DA, Manuel DG, Gunraj N, Anderson G, Naylor CD, Laupacis A. Age, risk-benefit trade-offs, and the projected effects of evidence-based therapies. Am J Med. 2004 Apr 15;116(8):540-5. doi: 10.1016/j.amjmed.2003.10.039. PMID 15063816
- [Result] Tinetti ME, Bogardus ST Jr, Agostini JV. Potential pitfalls of disease-specific guidelines for patients with multiple conditions. N Engl J Med. 2004 Dec 30;351(27):2870-4. doi: 10.1056/NEJMsb042458. No abstract available. PMID 15625341
- [Result] Tegn N, Abdelnoor M, Aaberge L, Endresen K, Smith P, Aakhus S, Gjertsen E, Dahl-Hofseth O, Ranhoff AH, Gullestad L, Bendz B; After Eighty study investigators. Invasive versus conservative strategy in patients aged 80 years or older with non-ST-elevation myocardial infarction or unstable angina pectoris (After Eighty study): an open-label randomised controlled trial. Lancet. 2016 Mar 12;387(10023):1057-1065. doi: 10.1016/S0140-6736(15)01166-6. Epub 2016 Jan 13. PMID 26794722
- [Result] Seto TB, Taira DA, Berezin R, Chauhan MS, Cutlip DE, Ho KK, Kuntz RE, Cohen DJ. Percutaneous coronary revascularization in elderly patients: impact on functional status and quality of life. Ann Intern Med. 2000 Jun 20;132(12):955-8. doi: 10.7326/0003-4819-132-12-200006200-00005. PMID 10858178
- [Result] Chait R, Zad O, Ramineni R, Shukla A, Mitchell A. Midterm outcomes and quality of life following percutaneous coronary intervention in nonagenarians. Am J Cardiol. 2011 Jun 1;107(11):1609-12. doi: 10.1016/j.amjcard.2011.01.046. Epub 2011 Mar 21. PMID 21420046
- [Result] Patel A, Rendu A, Moran P, Leese M, Mann A, Knapp M. A comparison of two methods of collecting economic data in primary care. Fam Pract. 2005 Jun;22(3):323-7. doi: 10.1093/fampra/cmi027. Epub 2005 Apr 11. PMID 15824056
- [Result] Caro JJ, Briggs AH, Siebert U, Kuntz KM; ISPOR-SMDM Modeling Good Research Practices Task Force. Modeling good research practices--overview: a report of the ISPOR-SMDM Modeling Good Research Practices Task Force--1. Value Health. 2012 Sep-Oct;15(6):796-803. doi: 10.1016/j.jval.2012.06.012. PMID 22999128
- [Result] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Result] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Result] TRIUMPH Investigators; Alexander JH, Reynolds HR, Stebbins AL, Dzavik V, Harrington RA, Van de Werf F, Hochman JS. Effect of tilarginine acetate in patients with acute myocardial infarction and cardiogenic shock: the TRIUMPH randomized controlled trial. JAMA. 2007 Apr 18;297(15):1657-66. doi: 10.1001/jama.297.15.joc70035. Epub 2007 Mar 26. PMID 17387132
- [Result] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- See also: Organisation WH. — http://www.who.int/healthinfo/survey/ageingdefnolder/en/